CLINICAL TRIAL: NCT06812078
Title: A Dose-Finding, Adaptive, Randomized, Double-Blinded, Placebo-Controlled Trial to Evaluate the Safety, Tolerability, and Efficacy of TAK-360 in Participants With Idiopathic Hypersomnia (IH)
Brief Title: A Study of TAK-360 in Adults With Idiopathic Hypersomnia
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TAK-360-2002; 2024-517712-29-00 (EU CTIS Number); jRCT2031240669 (Registry Identifier: jRCT)
Record Dates: First submitted 2025-02-03; First posted 2025-02-06 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: Idiopathic Hypersomnia
Keywords: Idiopathic Hypersomnia; TAK-360
MeSH Terms: conditions — Idiopathic Hypersomnia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- TAK-360 (Experimental): Participants will receive TAK-360 tablets, orally, for 4 weeks.
  Interventions: Drug: TAK-360
- Placebo (Placebo Comparator): Participants will receive TAK-360 matching placebo tablets, orally, for 4 weeks.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: TAK-360 — TAK-360 tablet.
  Arms: TAK-360
Other: Placebo — TAK-360 matching placebo tablet.
  Arms: Placebo

SUMMARY:
Idiopathic Hypersomnia (IH) is a condition where people feel extremely sleepy during the day, especially in the morning, even if they sleep a lot at night. They may have trouble waking up in the morning, no matter how much they sleep (sometimes more than 11 hours per day), and they can't help feeling tired, even after taking daytime naps. Because of this sleepiness, they may have trouble focusing, thinking clearly, or keeping up with daily activities. They may also have symptoms like dizziness or feeling lightheaded. Orexin is a chemical made in the brain that helps keep a person awake and alert. TAK-360 acts like orexin. Previous studies have shown that medicines that act like orexin may keep people awake.

The main aim of this study is to learn how safe TAK-360 is and how well adults with IH tolerate it. Researchers also want to find out if TAK-360 can help people with IH stay awake and how much TAK-360 is needed to do that.

Participants will be randomly (by chance, like drawing names from a hat) chosen to receive either TAK-360 or a placebo. The placebo looks just like TAK-360 but does not have any medicine in it. Using a placebo helps researchers learn about the real effect of the treatment.

ELIGIBILITY:
Key Inclusion Criteria:

1. The participant weighs greater than or equal to (≥) 40 kilograms (kg) and has a body mass index (BMI) between 16 and 38 kilograms per meter square (kg/m^2) [inclusive].
2. The participant has a documented, current diagnosis of IH.

Key Exclusion Criteria:

1. The participant has a current medical disorder associated with excessive daytime sleepiness (EDS) [other than IH].
2. The participant has medically significant thyroid disease.
3. The participant has a history of cancer in the past 5 years. (This exclusion does not apply to participants with carcinoma in situ [such as basal cell carcinoma] that has been treated and is stable, or who have been stable without further treatment. These participants may be included after approval by the medical monitor.)
4. The participant has any of the following viral infections based on a positive test result: Hepatitis B surface antigen (at screening), hepatitis C virus antibody (at screening), human immunodeficiency virus (HIV) antibody/antigen (at screening).
5. The participant has a clinically significant history of head injury or head trauma.
6. The participant has history of epilepsy, seizure, or convulsion (exception for a single febrile seizure in childhood).
7. The participant has a history of cerebral ischemia, transient ischemic attack (less than [<]5 years from screening), intracranial aneurysm, or arteriovenous malformation.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Estimated)
Dates: Start 2025-02-07 (Actual); Primary Completion 2026-07-16 (Estimated); Study Completion 2026-07-16 (Estimated)

PRIMARY OUTCOMES:
Number of Participants With at Least One Treatment-emergent Adverse Events (TEAEs) | Up to Week 8
  An adverse event (AE) is any untoward medical occurrence in a clinical investigation participant administered a pharmaceutical product. A TEAE is defined as any event emerging or manifesting at or after the initiation of treatment with a study intervention or medicinal product or any existing event that worsens in either intensity or frequency following exposure to the study intervention or medicinal product.

SECONDARY OUTCOMES:
Change from Baseline at Week 4 in Epworth Sleepiness Scale (ESS) Total Score | Baseline, Week 4
  The ESS provides individuals with 8 different situations of daily life and asks them how likely they are to fall asleep in those situations (scored 0 to 3) and to try to imagine their likelihood of dozing even if they have not actually been in the identical situation; the scores are summed to give an overall score of 0 to 24. Higher scores indicate stronger subjective daytime sleepiness, and scores below 10 are considered to be within the normal range.
Change from Baseline at Week 4 in Idiopathic Hypersomnia Severity Scale (IHSS) Total Score | Baseline, Week 4
  IHSS is a 14-item self-assessment questionnaire, to measure the severity, frequency and functional impact of the three key IH symptoms (during a recall period of "past 7 days"). The IHSS includes 14 items in total; two items (1 and 2) on nighttime sleep duration and quality, three items (3, 4 and 5) on sleep inertia and sleep drunkenness after nighttime sleep and one (8) after daytime nap, and three items (6, 7 and 9) on diurnal symptoms (nap occurrence, daytime sleepiness). Items 10 to 14 assess daytime functioning alterations due to hypersomnolence. Six items are scored on a 3-point Likert scale and eight items on a 4-point Likert scale; the Likert scale is a point scale which is used to allow the individual to express how much they agree or disagree with a particular statement. The total IHSS score is the sum of all item scores (range: 0 to 50), and higher scores indicate more severe symptoms.

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (29):
- United States (13):
  - Takeda Site 11, Redwood City, California
  - Takeda Site 10, Santa Ana, California
  - Takeda Site 27, Colorado Springs, Colorado
  - Takeda Site 19, Brandon, Florida
  - Takeda Site 14, Winter Park, Florida
  - Takeda Site 29, St Louis, Missouri
  - Takeda Site 16, Denver, North Carolina
  - Takeda Site 15, Huntersville, North Carolina
  - Takeda Site 12, Cincinnati, Ohio
  - Takeda Site 17, Cincinnati, Ohio
  - Takeda Site 13, Columbia, South Carolina
  - Takeda Site 18, San Antonio, Texas
  - Takeda Site 28, Norfolk, Virginia
- France (3):
  - Takeda Site 1, Montpellier, Hrault
  - Takeda Site 3, Nantes, Pays de Loire
  - Takeda Site 2, Paris
- Takeda Site 4, Shatin, Hong Kong
- Italy (4):
  - Takeda Site 6, Pozzilli, Isernia
  - Takeda Site 7, Rome, Roma
  - Takeda Site 26, Verona, Veneto
  - Takeda Site 5, Bologna
- Japan (6):
  - Takeda Site 25, Fukuoka-Shi Hakata-Ku, Fukuoka
  - Takeda Site 23, Kurume-shi, Fukuoka
  - Takeda Site 22, Kohoku-ku, Yokohama-Shi, Kanagawa
  - Takeda Site 20, Kumamoto, Kumamoto
  - Takeda Site 21, Yodogawa-ku, Osaka-shi, Osaka
  - Takeda Site 24, Bunkyo-ku, Tokyo
- Spain (2):
  - Takeda Site 9, Vitoria-Gasteiz, Alava
  - Takeda Site 8, Madrid

IPD SHARING:
Plan to Share IPD: Yes
Takeda provides access to the de-identified individual participant data (IPD) for eligible studies to aid qualified researchers in addressing legitimate scientific objectives (Takeda's data sharing commitment is available on https://clinicaltrials.takeda.com/takedas-commitment?commitment=5). These IPDs will be provided in a secure research environment following approval of a data sharing request, and under the terms of a data sharing agreement.
Supporting Information: Study Protocol, SAP, ICF, CSR
Access Criteria: IPD from eligible studies will be shared with qualified researchers according to the criteria and process described on https://vivli.org/ourmember/takeda/. For approved requests, the researchers will be provided access to anonymized data (to respect patient privacy in line with applicable laws and regulations) and with information necessary to address the research objectives under the terms of a data sharing agreement.
URL: https://vivli.org/ourmember/takeda/

REFERENCES:
- See also: Click here for more information about this trial in easy-to-understand language, including a Plain Language Summary of the results if the trial has been completed. — https://clinicaltrials.takeda.com/study-detail/88ad04fc158b4d5a??page=1&idFilter=TAK-360-2002